CLINICAL TRIAL: NCT01564550
Title: The Effect of Type 2 Diabetes and Dietary Regulation on VLDL1-and VLDL2-triglyceride Metabolism
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 33046
Record Dates: First submitted 2012-02-22; First posted 2012-03-28 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2012-11

CONDITIONS: Type 2 Diabetes; Dyslipidemia
Keywords: Type 2 diabetes; Very-low-density-lipoprotein(VLDL); VLDL1; VLDL2; hyperinsulinemia; diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias; Hyperinsulinism | interventions — Insulin; Diet

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- type 2 diabetes
  Interventions: Drug: Insulin
- healthy subjects
  Interventions: Drug: insulin; Other: diet; Other: no diet

INTERVENTIONS:
Drug: Insulin — Insulin is given as a constant infusion( 0,6 mU/kg/min) during the hyperinsulinemia period of the study lasting four and a half hour.
  Other Names: Actrapid, Novo Nordisk, A10AB01
  Groups: type 2 diabetes
Drug: insulin — Insulin is given as a constant infusion( 0,6 mU/kg/min) during the hyperinsulinemia period of the study lasting four and a half hour.
  Other Names: Actrapid, Novo Nordisk, A10AB01
  Groups: healthy subjects
Other: diet — The subjects ingest a three day isocaloric diet (55 % carbohydrate,30% fat, 15 % protein)prior to the study day.
  Groups: healthy subjects
Other: no diet — The subjects will ingest a non-restricted diet prior to the study day.
  Groups: healthy subjects

SUMMARY:
In this study the investigators wish to compare Very Low-Density Lipoprotein (VLDL) kinetics in type 2 diabetic males and healthy males postabsorptive and during hyperinsulinemia. The kinetics is obtained using an ex-vivo VLDL1- and VLDL2-triglyceride labeling technique. The investigators hypothesis is that the investigators will find an increased VLDL1 production in type 2 diabetic males, which is not lowered by hyperinsulinemia. Also the investigators wish to investigate the influence of diet on VLDL1 and VLDL2 production in healthy males, where the investigators expect less variance in VLDL production when the subject is given an isocaloric diet.

DETAILED DESCRIPTION:
Patients with type 2 diabetes are more likely to suffer from dyslipidemia. Earlier research has shown that these patients have an increased VLDL production and this could be a key factor in dyslipidemia development. Especially the production of VLDL1 seems to be increased where an inhibitory response to insulin is lacking. Further investigation in VLDL1 and VLDL2 kinetics is required.

The investigators wish:

1. To extend the method of ex vivo labeling of VLDL-triglyceride, to include separate labeling of VLDL1- and VLDL2-triglyceride for evaluation of the separate lipoprotein subtype kinetics.
2. To investigate VLDL1- and VLDL2-triglyceride kinetics in the post absorptive state and under experimental hyperinsulinemia in twelve type 2 diabetic males compared to twelve healthy age, sex, and BMI matched males.
3. To investigate the effect of a three day isocaloric diet compared to a non-restricted diet on the day-to-day variation in VLDL1 and VLDL2-triglyceride kinetics in healthy men. The investigators here examine six subjects on two different days who ingest a non-restricted diet and compare this group to six subjects examined on two different days, who have prior ingest a three day isocaloric diet.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes during at least six month or healthy subjects
* male
* BMI 25-36 kg/m2
* age 35-65

Exclusion Criteria:

* other diseases (hypertension and hypercholesterolemia tolerated)
* Insulin treatment
* alcohol abuse
* smoking
* medication affecting lipid metabolism apart from statins and antihypertensive drugs paused 2 weeks prior to the study day.
* participation in studies involving radioactive isotopes or larger x-ray investigations within the last six month.
* blood donation within three month.

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The type 2 diabetic men will be recruited from the endocrinology ambulatory of Aarhus University hospital. The healthy subjects will be recruited by local advertisement in the city of Aarhus and by national website advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
VLDL1 and VLDL2-triglyceride secretion rate (µmol/min) | 7 hours
  VLDL1 and VLDL2 kinetics assessed over a single study day.

CONTACTS AND LOCATIONS:
Overall Officials: Rakel F Johansen, M.D., Principal Investigator — University of Aarhus
Locations (1):
- Department of Endocrinology MEA, Aarhus Hospital, Aarhus C, Denmark

REFERENCES:
- [Derived] Johansen RF, Sondergaard E, Sorensen LP, Jurik AG, Christiansen JS, Nielsen S. Basal and insulin-regulated VLDL1 and VLDL2 kinetics in men with type 2 diabetes. Diabetologia. 2016 Apr;59(4):833-43. doi: 10.1007/s00125-015-3856-5. Epub 2016 Jan 19. PMID 26781548